CLINICAL TRIAL: NCT04760587
Title: Application of Smart Devices in Adolescent Weight Control: A Longitudinal Panel Study
Brief Title: Application of Smart Devices in Adolescent Weight Control
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202005008RIND
Record Dates: First submitted 2021-02-17; First posted 2021-02-18 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2022-04

CONDITIONS: Adolescent Obesity
Keywords: Adolescent; smart devices; weight control; health literacy
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: smart devices in adolescent
  Interventions: Behavioral: smart devices in adolescent weight control

INTERVENTIONS:
Behavioral: smart devices in adolescent weight control — The study will apply mobile phone applications and smart watches to understand the relationship between weight control behaviors and weight control health outcome in adolescent.

SUMMARY:
According to the definition of Health Literacy, health literacy means that a person can apply his or her reading, writing, and computing abilities to health-related information and activities. WHO consider Health Literacy is the cognitive and social skills which determine the motivation and ability of individuals to gain access, to understand and use information.

The purposes of this study will to understand the relationship between health literacy, weight control behavior and weight control health outcome.

DETAILED DESCRIPTION:
According to the definition of Health Literacy, health literacy means that a person can apply his or her reading, writing, and computing abilities to health-related information and activities. WHO consider Health Literacy is the cognitive and social skills which determine the motivation and ability of individuals to gain access, to understand and use information.

The purposes of this study will to understand the relationship between health literacy, weight control behavior and weight control health outcome.

According to the purpose, the study will be multi wave longitudinal panel study. The study will apply mobile phone applications and smart watches to understand the relationship between weight control behaviors and weight control health outcome in adolescent.

There are two blocks in the mobile phone applications: questionnaire block and Weight status block will be design for the study. Questionnaire block include demography, and health literacy scales and diet diary. Weight status block include height, weight, waist circumference, and hip circumference. After the participant key-in the height and weight, the system will automatically calculate the BMI, also show the results of the BMI. The standard for BMI interpretation was by Dr. Chang's research about New Growth Charts for Taiwanese Adolescents.

The data of smart watches will be upload into the NTUH health cloud system (named NTU MED GOD). This is the NTUH health cloud, different kinds of medical materials and data could be sent to the system, such as mobile phone and smart watches data.

ELIGIBILITY:
Inclusion Criteria:

* 13-19 years old adolescents;
* Could use their mobile phones to upload diet records and fill out the questionnaire;
* Adolescents and their parents agree to involve in the study and sign the consent form.

Exclusion Criteria:

* Severe diseases;
* Participate in other weight control program.

Ages: 13 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study in this study will be 13-19 years old adolescents.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
BMI(body mass index) | Change from baseline body mass index at 3 months, 6 months, 9 months, and 12 months.
  Body mass index (BMI) is a measure of body fat based on height and weight.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsia Chen, Principal Investigator — National Taiwan University, College of Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No